CLINICAL TRIAL: NCT03103789
Title: Assessment of Esophageal Epithelium Integrity With Use of a Novel Mucosal Impedance Device
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Sandhill Scientific (Industry)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 140470
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GERD patients: Patients who are undergoing standard of care EGD with or without BRAVO pH capsule placement and have been diagnosed with GERD will have mucosal impedance measured by single catheter and balloon assembly.
  Interventions: Diagnostic Test: single catheter mucosal impedance testing; Diagnostic Test: balloon assembly mucosal impedance testing
- control: Patients who are undergoing standard of care EGD with or without BRAVO pH capsule placement will have mucosal impedance measured by single catheter and balloon assembly.
  Interventions: Diagnostic Test: single catheter mucosal impedance testing; Diagnostic Test: balloon assembly mucosal impedance testing

INTERVENTIONS:
Diagnostic Test: single catheter mucosal impedance testing
Diagnostic Test: balloon assembly mucosal impedance testing

SUMMARY:
The objective of this study is to design and use a novel, minimally invasive mucosal impedance (MI) technology to inexpensively and accurately test mucosal health in suspected gastroesophageal reflux disease (GERD) and nonerosive reflux disease (NERD) patients as compared to those without GERD.

DETAILED DESCRIPTION:
During routine esophagogastroduodenoscopy (EGD), consented study participants will have the original single channel MI catheter advanced through the working channel of the endoscope. Measurements will be taken at 3 locations for 5 seconds each. The catheter will then be removed and a custom-designed balloon assembly will be inserted through the working channel of the endoscope. The balloon assembly will expand to a maximum diameter of 2 cm spanning from the distal to mid esophagus and contain external metal contacts to form 40 impedance channels made up by 10 axial channels spanning a 10 cm axial area and four radial channels.This design will allow us to measure mucosal impedance both axially and radially thus enabling us to assess the discriminating ability of the device for reflux disease. The balloon assembly will be held in place for 5 seconds. Once the mucosal impedance data have been recorded, the balloon assembly will be deflated and removed by the investigator. The study procedure will add approximately 1-3 minutes of procedure time for each research participant.

Those participants who are diagnosed with Grade C or D esophagitis at the initial visit will return for a follow-up visit after treatment with proton pump inhibitor (PPI) therapy to determine whether or not esophagitis has healed as part of their standard of care. If no esophagitis is detected at the follow-up EGD, we will gather one final comparison MI reading during this visit. If esophagitis is still present, follow-up MI will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing standard of care EGD with or without BRAVO pH capsule placement

Exclusion Criteria:

* Age less than 18 years old
* Patients unable to give informed consent
* Use of acid suppressive therapy within last 10 days
* Known history of Barrett's esophagus or gastric surgery, other than non-functioning (slipped) Nissen fundoplication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for endoscopic procedures (esophagogastroduodenoscopy (EGD)) by the principal investigator as part of their routine care and who do not meet any of the pre-defined exclusion criteria will be considered for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2014-04-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
mucosal impedance values | Values will be obtained at conclusion of EGD, an expected average of 6 minutes
  compare the mucosal impedance values obtained from single channel catheter and balloon assembly catheter in GERD patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel DA, Higginbotham T, Slaughter JC, Aslam M, Yuksel E, Katzka D, Gyawali CP, Mashi M, Pandolfino J, Vaezi MF. Development and Validation of a Mucosal Impedance Contour Analysis System to Distinguish Esophageal Disorders. Gastroenterology. 2019 May;156(6):1617-1626.e1. doi: 10.1053/j.gastro.2019.01.253. Epub 2019 Jan 31. PMID 30711626